CLINICAL TRIAL: NCT06080503
Title: G-FORCE: Phase II Randomized Study of Glottic Larynx Hypofractionated Radiotherapy Versus ConvEntional Radiotherapy
Brief Title: Phase II Randomized Study of Hypofractionated Versus Conventional Radiotherapy
Acronym: G-FORCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, David Sher, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0715
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Laryngeal Carcinoma
Keywords: Larynx
MeSH Terms: conditions — Laryngeal Neoplasms; Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Highly conformal hypofractionated radiotherapy (Experimental): LT-SABR 42.5 Gy in 5 fractions Low-risk: twice/week Moderate-risk: weekly
  Interventions: Radiation: LT-SABR
- Conventional radiotherapy (Experimental): Conventional Radiotherapy 63 Gy in 28 fractions (T1) 65.25 Gy in 29 fractions (T2)
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: LT-SABR — 42.5 Gy in 5 fractions Low-risk: twice/week Moderate-risk: weekly
  Arms: Highly conformal hypofractionated radiotherapy
Radiation: IMRT — 63 Gy in 28 fractions (T1) 65.25 Gy in 29 fractions (T2)
  Arms: Conventional radiotherapy

SUMMARY:
To compare the acute tolerance of highly conformal hypofractionated versus conventional radiotherapy.

DETAILED DESCRIPTION:
Screening/Baseline Procedures Assessments performed exclusively to determine eligibility for this study will be done only after obtaining informed consent. Assessments performed for clinical indications (not exclusively to determine study eligibility) may be used for baseline values even if the studies were done before informed consent was obtained.

All screening procedures must be performed within 30 days prior to registration into the study unless otherwise stated. The screening procedures include:

Informed Consent Medical history--Complete medical and surgical history Demographics--Age, gender, race, ethnicity Review subject eligibility criteria Review previous and concomitant medications Physical exam including vital signs, height and weight Vital signs (temperature, pulse, respirations, blood pressure), height, weight Performance status--Performance status evaluated prior to study entry. If there is any variability in the physicians' notes, the higher number will be used for research purposes.

Positron emission tomography-computerized tomography or computerized tomography of neck (any time prior to registration) Laryngoscopy Pregnancy test (for females of child-bearing potential) Quality of life Questionnaires and Symptom Questionnaires --EORTC QLQ-C30, H&N 35, VHI, and EQ-5D. These forms will be referred to collectively as QoL Questionnaires. Can be given on paper, over the phone, or in EPIC as needed.

Procedures During Treatment Day 1-First fraction of radiotherapy per standard, departmental stereotactic protocol

Follow-up Procedures--After initial follow-up at 2 weeks (+/- 7 days) after completion of radiation therapy, subjects will be followed at 3 months and 12 months. These protocol mandated procedures will occur at each follow-up:

Interim history Physical exam, vital signs, ECOG Performance Status Laryngoscopy (optional at 1-2 weeks) to assess tumor response and toxicity Quality of life and voice quality assessment. Can be given on paper, over the phone, or in EPIC as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically-proven diagnosis of squamous cell carcinoma in situ, squamous cell carcinoma, or squamous cell variants (sarcomatoid, verrucous, basaloid, and papillary subtypes) involving the glottic larynx.
2. Clinical stage 0-II (AJCC, 8th edition) with direct laryngoscopy showing no evidence of greater than stage II true glottic larynx cancer and PET/CT or CT neck showing no evidence of regional disease.
3. Minimum age is 18 years.
4. ECOG Performance Status 0-2
5. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   5.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
6. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. AJCC stage III or stage IV larynx cancer
2. Involvement of the arytenoid cartilage beyond the vocal process.
3. Prior chemotherapy for treatment of the targeted larynx lesion.
4. Synchronous primaries in the head and neck
5. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation fields.
6. Subjects smoking in excess of 1 pack of cigarettes per day.
7. Subjects may not be receiving any other investigational agents.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-03-14 (Estimated)

PRIMARY OUTCOMES:
To compare the acute toxicity outcomes between patients treated with highly-conformal hypofractionated radiotherapy and conventional radiotherapy. | 3 months following treatment
  Acute toxicity score (i.e. T score), defined as the mean number of grade 2 or higher acute toxicities experienced between the start of radiotherapy and 3 months following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David Sher, MD, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States